CLINICAL TRIAL: NCT03228862
Title: Optimal Initial and Maintenance Doses of Ergocalciferol Supplementation for Treatment of Hypovitaminosis D in Thai Adults: A Randomized, Double-blinded Dose-comparison Study
Brief Title: Optimal Doses of Ergocalciferol Supplementation for Treatment of Hypovitaminosis D in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Lalita Wattanachanya, MD, Assist Prof., Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 088/60
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Vitamin D2 Supplementation in Vitamin D Insufficiency
MeSH Terms: interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- D40000 (Experimental): Patients are randomly assigned to receive Ergocalciferol 40000 IU once weekly
  Interventions: Drug: Ergocalciferol
- D60000 (Experimental): Patients are randomly assigned to receive Ergocalciferol 60000 IU once weekly
  Interventions: Drug: Ergocalciferol
- D80000 (Experimental): Patients are randomly assigned to receive Ergocalciferol 80000 IU once weekly
  Interventions: Drug: Ergocalciferol

INTERVENTIONS:
Drug: Ergocalciferol — Ergocalciferol 40000, 60000 and 80000 once weekly

SUMMARY:
To investigate the optimal initial and maintenance doses of vitamin D2 supplementation for the treatment of vitamin D insufficiency in Thai adults, and to determine the prevalence of and risk factors for hypovitaminosis D among Thai adults.

DETAILED DESCRIPTION:
A double-blinded prospective, randomized study undertaken at outpatient clinic of King Chulalongkorn Memorial Hospital. The patients with vitamin D insufficiency were included and divided into three groups according to their initial 25OHD concentrations. Patients are randomly assigned to receive vitamin D2 40000, 60000 or 80000 IU once weekly. Serum 25(OH)D levels are measured at 12 weeks after vitamin D2 supplemetaiton. The patients with 25OHD more than 30ng/mL are enroll into the maintenance phase of the study and are randomly assigned to receive vitamin D2 20000 or 40000 IU once weekly for another 12 months. The 25OHD concentration are measure again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age ≥ 15 years
2. BMI 18 - 35 kg/m2
3. Serum 25(OH)D < 30ng/ml

Exclusion Criteria:

1. Hypercalcemia, nephrolithiasis, or fractures
2. Hepatic disease
3. Kidney disease
4. Granulomatous disease
5. Currently supplemented with vitamin D

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
serum 25OHD phase 1 | 12 weeks
  serum 25OHD concentration after initial vitamin D2 supplemetaiton

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn Univerity and King Chulalongkorn Memorial Hospital, Bangkok, Thailand